CLINICAL TRIAL: NCT02676726
Title: STELLA 2 Trial: Staging of Endometrial and Ovarian Cancer Comparing the Transperitoneal vs. Extraperitoneal Approach for Laparoscopic Lymphadenectomy of Aortic Nodes, Evaluating Complications
Brief Title: STELLA 2 Trial: Transperitoneal vs. Extraperitoneal Approach for Laparoscopic Staging of Endometrial/Ovarian Cancer
Acronym: STELLA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P14/1817
Record Dates: First submitted 2015-10-14; First posted 2016-02-08 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Endometrial Neoplasms; Ovarian Neoplasms
Keywords: extraperitoneal; transperitoneal; laparoscopic aortic lymphadenectomy; endometrial cancer; ovarian cancer; surgical staging
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extraperitoneal (Experimental): Patients who where randomized to extraperitoneal laparoscopic aortic lymphadenectomy.
  Interventions: Procedure: Extraperitoneal Laparoscopic aortic lymphadenectomy
- Transperitoneal (Active Comparator): Patients who where randomized to transperitoneal laparoscopic aortic lymphadenectomy.
  Interventions: Procedure: Transperitoneal Laparoscopic aortic lymphadenectomy

INTERVENTIONS:
Procedure: Extraperitoneal Laparoscopic aortic lymphadenectomy — Aortic/para-aortic lymph nodes dissection and retrieval by extraperitoneal laparoscopy; the intervention may be completed by robotic-assisted or traditional laparoscopy.
  Other Names: Extraperitoneal laparoscopic para-aortic lymphadenectomy; Retroperitoneal laparoscopic lumbo-aortic lymphadenectomy
  Arms: Extraperitoneal
Procedure: Transperitoneal Laparoscopic aortic lymphadenectomy — Aortic/para-aortic lymph nodes dissection and retrieval by transperitoneal laparoscopy; the intervention may be completed by robotic-assisted or traditional laparoscopy.
  Other Names: Transperitoneal laparoscopic para-aortic lymphadenectomy; Transperitoneal laparoscopic lumbo-aortic lymphadenectomy
  Arms: Transperitoneal

SUMMARY:
The purpose of this study is to determine whether or not there are more complications in the extraperitoneal compared with the transperitoneal approach for laparoscopic aortic lymphadenectomy for the surgical staging of endometrial or ovarian cancer

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometrial cancer confirmed by histopathological analysis (endometrial biopsy) requiring surgical staging according to FIGO (the International Federation of Gynecology and Obstetrics) recommendations
* Diagnosis of ovarian cancer confirmed by histopathological analysis after an initial cystectomy or oophorectomy without suspicion of neoplasia thus requiring additional surgical staging according to FIGO recommendations

Exclusion Criteria:

* Diagnosis of advanced endometrial cancer based on findings on imaging techniques (CT, MRI and/or PET)
* Diagnosis of advanced endometrial or ovarian cancer based on intraoperative findings (e.g. peritoneal carcinomatosis at initial laparoscopy)
* Patients who underwent previous aortic lymphadenectomy
* Patients who received previous pelvic and/or aortic radiotherapy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09-08 (Actual)

PRIMARY OUTCOMES:
Surgical complications | intraoperatively, within 30 days after surgery, and past 30 days after surgery up to 3 months after surgery
  Composite outcome defined by including at least one of the following:
  * Total estimated blood loss > 500 mL during surgery
  * Blood transfusion
  * Intraoperative complication classified as Dindo grade III or worse, related to the aortic lymphadenectomy
  * Early postoperative complication (within 30 days after surgery) classified as Dindo grade III or worse, related to the aortic lymphadenectomy
  * Late postoperative complication (past 30 days after surgery) classified as Dindo grade III or worse, related to the aortic lymphadenectomy
  * Conversion to laparotomy during the aortic lymphadenectomy
  * Inability to complete the aortic lymphadenectomy

SECONDARY OUTCOMES:
Number of lymph nodes | Postoperatively (within 1 week), at the moment of histopathologic examination
  The number of lymph nodes (absolute number) is specified by the pathologist on histopathological analysis of the sample sent by the surgeon after surgical staging is realized (laparoscopic aortic lymphadenectomy). This variable is subdivided into: supra-mesenteric and infra-mesenteric.
Operative time | At the time of the surgery
  Total duration of surgery (from initial skin incision to end of skin suture), and total aortic lymphadenectomy time (time spent since the beginning of aortic lymphadenectomy to its completion). Metric: minutes.
Hospital stay | Measured the day the patient is discharged (up to 100 days)
  The number of days that patients stay in the hospital after surgery, measured in days from the day of the surgery to the day the patient is discharged from the hospital.
Overall survival | up to 3 years after surgery
  Number of patients alive after surgery.
Disease-free survival | up to 3 years after surgery
  Period of time in which there is no appearance of the symptoms or effects of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil Moreno, MD, PhD, Study Chair — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Berta Diaz Feijoo, MD, PhD, Study Director — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Alejandro Correa Paris, MD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; M. Assumpció Pérez-Benavente, MD, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Silvia Franco Camps, MD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Jose Luis Sánchez Iglesias, MD, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Silvia Cabrera Díaz, MD, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Oriol Puig Puig, MD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Javier De La Torre, MD, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona
Locations (1):
- Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Vasilev SA, McGonigle KF. Extraperitoneal laparoscopic para-aortic lymph node dissection. Gynecol Oncol. 1996 Jun;61(3):315-20. doi: 10.1006/gyno.1996.0149. PMID 8641608
- [Background] Dowdy SC, Aletti G, Cliby WA, Podratz KC, Mariani A. Extra-peritoneal laparoscopic para-aortic lymphadenectomy--a prospective cohort study of 293 patients with endometrial cancer. Gynecol Oncol. 2008 Dec;111(3):418-24. doi: 10.1016/j.ygyno.2008.08.021. Epub 2008 Oct 2. PMID 18835020
- [Background] Gil-Moreno A, Maffuz A, Diaz-Feijoo B, Puig O, Martinez-Palones JM, Perez A, Garcia A, Xercavins J. Modified approach for extraperitoneal laparoscopic staging for locally advanced cervical cancer. J Exp Clin Cancer Res. 2007 Dec;26(4):451-8. PMID 18365538
- [Background] Gil-Moreno A, Diaz-Feijoo B, Morchon S, Xercavins J. Analysis of survival after laparoscopic-assisted vaginal hysterectomy compared with the conventional abdominal approach for early-stage endometrial carcinoma: a review of the literature. J Minim Invasive Gynecol. 2006 Jan-Feb;13(1):26-35. doi: 10.1016/j.jmig.2005.08.013. PMID 16431320
- [Background] Gil-Moreno A, Diaz-Feijoo B, Perez-Benavente A, del Campo JM, Xercavins J, Martinez-Palones JM. Impact of extraperitoneal lymphadenectomy on treatment and survival in patients with locally advanced cervical cancer. Gynecol Oncol. 2008 Sep;110(3 Suppl 2):S33-5. doi: 10.1016/j.ygyno.2008.03.024. Epub 2008 Jun 5. PMID 18538379
- [Background] Gil-Moreno A, Franco-Camps S, Diaz-Feijoo B, Perez-Benavente A, Martinez-Palones JM, Del Campo JM, Parera M, Verges R, Castellvi J, Xercavins J. Usefulness of extraperitoneal laparoscopic paraaortic lymphadenectomy for lymph node recurrence in gynecologic malignancy. Acta Obstet Gynecol Scand. 2008;87(7):723-30. doi: 10.1080/00016340802136343. PMID 18607826
- [Background] Pakish J, Soliman PT, Frumovitz M, Westin SN, Schmeler KM, Reis RD, Munsell MF, Ramirez PT. A comparison of extraperitoneal versus transperitoneal laparoscopic or robotic para-aortic lymphadenectomy for staging of endometrial carcinoma. Gynecol Oncol. 2014 Feb;132(2):366-71. doi: 10.1016/j.ygyno.2013.12.019. Epub 2013 Dec 20. PMID 24361579
- [Background] Dowdy SC, Mariani A. Lymphadenectomy in endometrial cancer: when, not if. Lancet. 2010 Apr 3;375(9721):1138-40. doi: 10.1016/S0140-6736(09)62068-7. Epub 2010 Feb 24. No abstract available. PMID 20188409
- [Background] Mariani A, Dowdy SC, Cliby WA, Gostout BS, Jones MB, Wilson TO, Podratz KC. Prospective assessment of lymphatic dissemination in endometrial cancer: a paradigm shift in surgical staging. Gynecol Oncol. 2008 Apr;109(1):11-8. doi: 10.1016/j.ygyno.2008.01.023. Epub 2008 Mar 4. PMID 18304622
- [Background] Gil-Moreno A, Franco-Camps S, Cabrera S, Perez-Benavente A, Martinez-Gomez X, Garcia A, Xercavins J. Pretherapeutic extraperitoneal laparoscopic staging of bulky or locally advanced cervical cancer. Ann Surg Oncol. 2011 Feb;18(2):482-9. doi: 10.1245/s10434-010-1320-9. Epub 2010 Sep 14. PMID 20839058
- [Background] Diaz-Feijoo B, Gil-Ibanez B, Perez-Benavente A, Martinez-Gomez X, Colas E, Sanchez-Iglesias JL, Cabrera-Diaz S, Puig-Puig O, Magrina JF, Gil-Moreno A. Comparison of robotic-assisted vs conventional laparoscopy for extraperitoneal paraaortic lymphadenectomy. Gynecol Oncol. 2014 Jan;132(1):98-101. doi: 10.1016/j.ygyno.2013.11.004. Epub 2013 Nov 11. PMID 24231134
- [Derived] Bebia V, Gil-Moreno A, Hernandez A, Gilabert-Estelles J, Franco-Camps S, de la Torre J, Siegrist J, Chipirliu A, Cabrera S, Bradbury M, Perez-Benavente A, Diaz-Feijoo B. Robot-assisted Extraperitoneal Para-aortic Lymphadenectomy Is Associated with Fewer Surgical Complications: A Post Hoc Analysis of the STELLA-2 Randomized Trial. J Minim Invasive Gynecol. 2021 Dec;28(12):2004-2012.e1. doi: 10.1016/j.jmig.2021.05.009. Epub 2021 May 20. PMID 34022445
- [Derived] Diaz-Feijoo B, Bebia V, Hernandez A, Gilabert-Estalles J, Franco-Camps S, de la Torre J, Segrist J, Chipirliu A, Cabrera S, Perez-Benavente A, Gil-Moreno A. Surgical complications comparing extraperitoneal vs transperitoneal laparoscopic aortic staging in early stage ovarian and endometrial cancer. Gynecol Oncol. 2021 Jan;160(1):83-90. doi: 10.1016/j.ygyno.2020.10.038. Epub 2020 Nov 5. PMID 33160695